CLINICAL TRIAL: NCT02318875
Title: Investigation of Kritech Efficacy on Subjects Having Functional Discomfort Associated to Joints and Muscles Disorders
Acronym: Easykrill
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vivatech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-A00320-41/1
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: Inflammation; swell; pain; functional impairment; stiffness
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kritech group (Experimental): Subjects take 1 Kritech capsule per day (dose of 300mg)
  Interventions: Dietary Supplement: Kritech administration
- Placebo group (Placebo Comparator): Subjects take 1 placebo capsule per day
  Interventions: Other: Placebo adminstration

INTERVENTIONS:
Dietary Supplement: Kritech administration — 300mg/day (1 capsule) during 12 weeks; oral ingestion
  Arms: Kritech group
Other: Placebo adminstration — 1 placebo capsule per day during 12 weeks; oral ingestion
  Arms: Placebo group

SUMMARY:
Joints and muscles disorders are common symptoms in the population. They are characterized by swelling, pain, functional impairment and morning stiffness. These disorders can be really disabling and painful, affecting the person's quality life. The purpose of this clinical trial is to test Kritech (Krill oil) efficacy in reducing these symptoms in 154 subjects complaining functional discomfort associated to joints and muscles disorders.

DETAILED DESCRIPTION:
Epidemiological studies on prevalence and incidence of joints and muscles disorders are scares. Two epidemiological French studies recorded patients consulting their GP for widespread pain, whatever the cause. The most often cited pain localization was the musculoskeletal system (36-59% of the cases). In Europe the situation is similar, with arthritis and osteoarthritis representing the 42% of pains. According to the WHO (World Health Organization) the musculoskeletal system's disorders are the first cause of handicap in the worldwide population.

Krill oil is low in both saturated fatty acids and monounsaturated fatty acid and high in polyunsaturated fatty acid including a high proportion of (n-3) fatty acids and particularly EPA and DHA. There are strong evidences that krill oil may improve the comfort of sensitive joints thank to its n-3 fatty acids and phospholipids content. Particularly, after a supplementation with a dietary product containing pure krill oil, a reduction of systemic inflammation, trough reduction of CRP, was concomitantly accompanied by improvement of various clinical scores associated with joint flexibility, comfort and function. Despite this, there are no studies yet on healthy volunteers complaining the symptoms of rheumatologic pathologies, without being ill.

Here we performed a clinical trial on 154 subjects complaining functional discomfort associated to joints and muscles disorders. The principal objective was to test Kritech efficacy in reducing these symptoms.

Subjects were split in two groups, with one receiving Kritech and the second one the placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects;
* >18 years old;
* Complaining functional discomfort associated to joints and/or muscles disorders, motility disorders and/or initial SMFA score higher or equal to 15 ;
* Able to give a written or verbal informed consent,
* Affiliated or beneficiary of social security

Exclusion Criteria:

* IMC>30kg/m
* Acute or chronic, progressive joint disorders (arthrosis, rheumatoid arthritis, acute articular rheumatism) of first or second degree and correlated treatments;
* Subjects refusing of giving their written or verbal informed consent
* Subjects deprived of freedom following an administrative or judicial decision
* Participation to another clinical trial in the last four weeks;
* People who already participated to another research that comprises an exclusion period still ongoing at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
SMFA score | 12 weeks

SECONDARY OUTCOMES:
SMFA " dysfunction index " and " bother index " subscores | 12 weeks
MCS (Mental Composite Score) and PCS (Physical Composite Score) of SF-36® questionnaire | 12 weeks
Pain evaluated by EVA (Échelle Visuelle Analogique) | 12 weeks
Clinical Global Impression (CGI scale) | 12 weeks
Analgesics consumption | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Moore, Professor, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Plateforme de Recherche Clinique - CIC1401- Plurithématique Tripode 13A3 Hôpital PELLEGRIN, Bordeaux, France